CLINICAL TRIAL: NCT02628691
Title: Monitoring Liver Disease Progression in Hepatitis C/HIV Co-infected Patients With No-to-moderate Fibrosis, in Phnom Penh, Cambodia (HCV-Monitoring)
Brief Title: Monitoring Liver Disease Progression in Hepatitis C/HIV Co-infected Patients With No-to-moderate Fibrosis, in Phnom Penh, Cambodia
Acronym: HCV-Monitoring
Status: Terminated | Type: Observational
Why Stopped: All patients were started on HCV treatment
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Sihanouk Hospital Center of HOPE (Other); University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Other Study IDs: HCV-Monitoring
Record Dates: First submitted 2015-11-25; First posted 2015-12-11 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Hepatitis C; HIV
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Left over biological samples (whole blood plasma and serum)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HCV coinfection with no-to-moderate fibrosis
  Interventions: Other: Liver fibrosis progression

INTERVENTIONS:
Other: Liver fibrosis progression — A history taking and physical examination focused on hepatic disease and blood sampling for basic hematologic and hepatic function parameters will be performed. Patients will also be referred every year for ultrasound and transient elastography measurements and sampling for some additional liver function tests and measurement of HCV-RNA viral load.

SUMMARY:
Data on the progression of liver fibrosis in patients co-infected with HIV taking effective suppressive antiretroviral therapy with no fibrosis or mild-to-moderate fibrosis at baseline are scarce. This uncertainty is reflected in lack of clear guidance on the need for earlier (than F3-F4) treatment in co-infected patients.

Within our hepatitis C/HIV co-infection project in Cambodia, the investigators have the opportunity to monitor for short-term fibrosis progression in a cohort of co-infected patients with initial no-to-moderate fibrosis being identified during another ongoing study (HCV-Epi) and contribute relevant data to aid the risk/benefit analysis of postponing HCV treatment in HIV/HCV co-infected patients with initial fibrosis stage F0-F2.

The HCV-Monitoring study is a mono-centric prospective cohort study proposing a standardized follow-up (clinical, biological and imaging) to monitor for progression of hepatitis C disease in all patients with HIV infection (on anti-retroviral treatment or not) of Sihanouk Hospital Center of Hope (Phnom Penh, Cambodia) who have chronic HCV infection with GT-1, -2, -3 or -6 but are not considered in immediate need of HCV treatment.

All adult HIV-infected patients of the cohort (on ART or not yet on ART) of Sihanouk hospital Center of Hope who are identified during the HCV-Epi study having chronic HCV infection (all genotypes) and considered not in immediate need of HCV treatment (= Fibrosis stages F0-F2 and no clinical signs of extra-hepatic disease) will be considered for inclusion and invited to participate.

Approximately 70 HCV/HIV co-infected patients with no-to-moderate hepatic fibrosis will be enrolled in this study.

Beyond the baseline visit (HCV-Epi), follow-up visits are planned at 6, 12, 18 and 24 months. These patient visits will comprise of a history taking and physical examination focused on hepatic disease and blood sampling for basic hematologic and hepatic function parameters. Additionally, patients will be referred every year for ultrasound and transient elastography measurements and sampling for some additional liver function tests and measurement of HCV-RNA viral load.

DETAILED DESCRIPTION:
Data on the progression of liver fibrosis in patients co-infected with HIV taking effective suppressive antiretroviral therapy with no fibrosis or mild-to-moderate fibrosis at baseline are scarce. This uncertainty is reflected in lack of clear guidance on the need for earlier (than F3-F4) treatment in co-infected patients.

Within our hepatitis C/HIV co-infection project in Cambodia, the investigators have the opportunity to monitor for short-term fibrosis progression in a cohort of co-infected patients with initial no-to-moderate fibrosis being identified during another ongoing study (HCV-Epi) and contribute relevant data to aid the risk/benefit analysis of postponing HCV treatment in HIV/HCV co-infected patients with initial fibrosis stage F0-F2.

The HCV-Monitoring study is a mono-centric prospective cohort study proposing a standardized follow-up (clinical, biological and imaging) to monitor for progression of hepatitis C disease in all patients with HIV infection (on anti-retroviral treatment or not) of Sihanouk Hospital Center of Hope (Phnom Penh, Cambodia) who have chronic HCV infection with GT-1, -2, -3 or -6 but are not considered in immediate need of HCV treatment.

The study will be conducted in Sihanouk Hospital Center of Hope (SHCH) in Phnom Penh (Cambodia), more particularly within the ambulatory HIV clinic setting. SHCH is a non-governmental hospital providing comprehensive HIV care free of charge since March 2003, as part of the national antiretroviral (ARV) program. They dispose of an experienced HIV clinician, counselor and social worker team and several operational research studies were conducted within this setting.

All adult HIV-infected patients of the cohort (on ART or not yet on ART) of Sihanouk hospital Center of Hope who are identified during the HCV-Epi study having chronic HCV infection (all genotypes) and considered not in immediate need of HCV treatment (= Fibrosis stages F0-F2 and no clinical signs of extra-hepatic disease) will be considered for inclusion and invited to participate.

Approximately 70 HCV/HIV co-infected patients with no-to-moderate hepatic fibrosis will be enrolled in this study. No formal sample size is being calculated. The final sample will comprise all patients fulfilling the inclusion criteria.

The data collected from the HCV-Epi study will be considered as the baseline visit for the HCV-Monitoring study. Thereafter, visits are planned at 6, 12, 18 and 24 months follow-up. These patient visits will, beyond the habitual HIV follow-up, integrate a history taking and physical examination focused on hepatic disease and blood sampling for basic hematologic and hepatic function parameters. Additionally, patients will be referred every year for ultrasound and transient elastography measurements and sampling for some additional liver function tests and measurement of HCV-RNA viral load.

ELIGIBILITY:
Inclusion Criteria:

* Male and females
* ≥18 years
* Documented HIV infection
* Evidence of infection with hepatitis C virus (all genotypes): Positive anti-HCV antibody and HCV RNA
* Absence of advanced liver disease or clinical signs of extra-hepatic disease:

  * F0-F2 (< 9,5 kPa) established by transient elastography, and
  * No clinical signs of extra-hepatic disease
* Not on HCV antiviral treatment

Exclusion Criteria:

* Currently on/or history of hepatitis C treatment
* Patients with initial fibrosis stage ≥ F3 (≥ 9,5 kPA on transient elastography)
* Patients not able/willing to adhere to the consultation, laboratory and liver stiffness measurement testing schedule as proposed in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult HIV-infected patients of the SHCH cohort who have chronic HCV infection (all genotypes) with no-to-moderate hepatic fibrosis and not considered in immediate need of HCV treatment.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2015-12-17 (Actual); Primary Completion 2017-07-12 (Actual); Study Completion 2017-07-12 (Actual)

PRIMARY OUTCOMES:
Short-term progression to advanced liver fibrosis | 30 months
  Proportion of patients who progress to advanced liver fibrosis (F≥3; LSM ≥9.5 kPa).

SECONDARY OUTCOMES:
Demographic characteristics | Baseline
  Demographic baseline characteristics of the study participants
Clinical characteristics | Baseline
  Clinical baseline characteristics of the study participants
Laboratory characteristics | Baseline
  Laboratory baseline characteristics of the study participants
Progression to cirrhosis | 30 months
  Proportion of patients who progress to cirrhosis ((F=4, > 14 kPa)
Liver stiffness measurement | 30 months
  Median Liver stiffness measurement increase per year
Changes in fibrosis stage scores | 30 months
  Change in Metavir score (regression/progression, number of stages difference)
Diagnostic accuracy of non-invasive serum bio-markers: APRI | 30 months
  Predictive value of APRI to identify a shift from (≤F2) to advanced fibrosis (≥3)
Diagnostic accuracy of non-invasive serum bio-markers: FIB-4 | 30 months
  Predictive value of FIB-4 to identify a shift from (≤F2) to advanced fibrosis (≥3)
Predictive factors for liver fibrosis progression | 30 months
  Factors associated with rapid fibrosis progression in HCV/HIV coinfected patients with initial mild to moderate fibrosis: age, gender, alcohol use, smoking, coffee consumption, comorbidities, liver enzymes, HCV viral load, HIV viral load, and ART exposure

CONTACTS AND LOCATIONS:
Overall Officials: Anja De Weggheleire, MD, Study Director — Institute of Tropical Medicine, Antwerp, Belgium; An Sokkab, MD, Principal Investigator — Sihanouk Hospital Center of HOPE (SHCH), Cambodia
Locations (1):
- Sihanouk Hospital Center of HOPE (SHCH), Cambodia, Phnom Penh, Cambodia